CLINICAL TRIAL: NCT01854684
Title: A Phase I Study of Surgery Plus Intraoperative Photodynamic Therapy (PDT) With Temoporfin in Patients With Resectable Primary Non-small Cell Lung Cancer (NSCLC) With Ipsilateral Thoracic Nodal (N1 or N2) or T3/T4 Disease
Brief Title: Photodynamic Therapy During Surgery in Treating Patients With Non-small Cell Lung Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 228112; NCI-2013-00886 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 228112 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — temoporfin; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (surgery and intraoperative PDT) (Experimental): Patients receive temoporfin IV over no less than 6 minutes and then undergo standard surgical resection with intraoperative PDT.
  Interventions: Drug: Temoporfin; Procedure: Therapeutic Conventional Surgery; Drug: Photodynamic Therapy; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Temoporfin — Given IV
  Other Names: Foscan; mTHPC
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection
Drug: Photodynamic Therapy — Undergo intraoperative PDT
  Other Names: Light Infusion Therapy™; PDT; Photoradiation Therapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of photodynamic therapy during surgery in treating patients with non-small cell lung cancer that can be removed by surgery. Photodynamic therapy uses a drug, such as temoporfin, that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed. This may be a better way to treat patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that intraoperative adjuvant regional photodynamic therapy with low-dose temoporfin is safe.

SECONDARY OBJECTIVES:

I. Initial assessment of efficacy (i.e., 2-year disease free survival). II. To investigate the relationship between signal transducer and activator of transcription 3 (STAT3) levels, measured light dose and the clinical outcome.

III. Correlate the serum concentrations of vitamin D metabolites (25-hydroxyvitarnin D3 and 1,25-dihydroxyvitamin D3) with the presence of lymph node (LN) metastasis at the time of surgical resection.

IV. To measure temoporfin uptake in malignant and normal tissue.

OUTLINE: This is a dose-escalation study of photodynamic therapy with temoporfin.

Patients receive temoporfin intravenously (IV) over no less than 6 minutes and then undergo standard surgical resection with intraoperative photodynamic therapy (PDT).

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC)
* Patients with resectable primary NSCLC who are undergoing surgery to resect T3 to T4 lesions OR any patients with clinical NI or N2 disease regardless of T-stage
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) scale of 0-2
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 6 months after surgery; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* The subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent prior to receiving any study related procedure
* Must consent to participate in study I 03103: Roswell Park Cancer Institute (RPCI) Data Bank and Biorepository (DBBR)

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with known brain metastases should be excluded from this clinical trial
* Patients with porphyria, or with known hypersensitivity to porphyrins or porphyrin-like compounds
* White blood cell (WBC) < 4,000
* Platelet count < 100,000
* Total serum bilirubin > 2 mg/dL
* Serum creatinine > 2 mg/dL
* Alkaline phosphatase (hepatic) or serum glutamic oxaloacetic transaminase (SGOT) > 3 times the upper normal limit
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of PDT with temoporfin, defined as the dose level in which more than 1 of 6 patients experience a dose limiting toxicity using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4 | 2 weeks

SECONDARY OUTCOMES:
Locoregional recurrence-free rate | Up to 2 years
  Estimated using simple relative frequencies. The corresponding 95% confidence interval for the estimated probability will be computed using the method proposed by Clopper and Pearson. Maximum likelihood estimation will be utilized in the model fitting procedures.
Overall survival | Up to 2 years
  Distribution will be obtained using the Kaplan-Meier method. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed.
Progression free survival | Up to 2 years
  Distribution will be obtained using the Kaplan-Meier method. Corresponding confidence intervals using the methodology of Brookmeyer and Crowley will be computed.
Toxicity rate, using NCI CTCAE version 4 | Up to 30 days after completion of study treatment
  Estimated using simple relative frequencies. The corresponding 95% confidence interval for the estimated probability will be computed using the method proposed by Clopper and Pearson. Maximum likelihood estimation will be utilized in the model fitting procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Chukwumere Nwogu, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States